CLINICAL TRIAL: NCT03149848
Title: Phase I, Single-center, Open Label, Fixed-sequence Cross-over Study to Evaluate the Effect of Rifabutin on the Pharmacokinetics of Oral Cabotegravir in Healthy Subjects
Brief Title: Effect of Rifabutin on the Pharmacokinetics of Oral Cabotegravir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205712; 2017-000103-25 (EudraCT Number)
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2019-02-04 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: Tuberculosis; Human Immunodeficiency Virus; Rifabutin; Drug-drug interaction; Cabotegravir
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections; Tuberculosis | interventions — cabotegravir; Rifabutin

STUDY DESIGN:
Intervention Model Description: This is a 2-period crossover study in healthy adults
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will be administered a single oral dose of CAB 30 mg after an overnight fast of at least 6 hours for 14 days in Period 1. Dosing of study medication on non-PK days may be with or without food.
  Interventions: Drug: Cabotegravir
- Treatment B (Experimental): Participants will be administered a single dose of RBT 300 mg and a single dose of CAB 30 mg after an overnight fast of at least 6 hours once daily for 14 days in Period 2. Dosing of study medication on non-PK days may be with or without food.
  Interventions: Drug: Cabotegravir; Drug: Rifabutin

INTERVENTIONS:
Drug: Cabotegravir — It will be available as a white aquarius film coated tablet for oral administration. CAB Tablet is composed of GSK1265744B (micronized) lactose monohydrate, microcrystalline cellulose, hypromellose, sodium starch glycolate, magnesium stearate
Drug: Rifabutin — It will be available as an opaque red-brown hard gelatin capsules containing 150 mg of rifabutin for oral administration. These capsules are composed of rifabutin, microcrystalline cellulose, sodium lauryl sulphate, magnesium stearate, and silica gel
  Arms: Treatment B

SUMMARY:
This is a Phase I, single-center, open-label, fixed-sequence, 2-period crossover study in healthy adults to evaluate the effect of oral rifabutin (RBT) 300 milligram (mg) on the pharmacokinetics of oral cabotegravir (CAB) 30 milligram ( mg). This study will evaluate the drug-drug interaction (DDI) potential between CAB and RBT to inform dosing strategies for tuberculosis in subjects receiving CAB for human immunodeficiency virus (HIV) treatment or prevention. In Treatment Period 1 (Treatment A) participants will receive CAB 30 mg once daily for 14 days, followed by Treatment Period 2 (Treatment B) where participants will receive RBT 300 mg once daily with CAB 30 mg once daily for 14 days. The total study duration will be approximately for 10 weeks. Approximately 15 healthy subjects will be enrolled to ensure that 12 subjects complete dosing and critical assessments.

ELIGIBILITY:
Inclusion Criteria

* Males and females between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Additionally, laboratory assessments that are specifically listed in the inclusion or exclusion criteria and are outside of the reference range can be repeated once during the screening period.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 18.5 - 31.0 kg/ meter square (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test), not lactating, and if she is of:

  * Non-reproductive potential defined as pre-menopausal with documented tubal ligation, hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Bilateral Oophorectomy, Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause FSH: >40 milli international unit/mililiter (MIU/mL) and estradiol <40 picogram (pg)/mL (<147 picomoles/L) is confirmatory];
  * Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication until the completion of the follow-up visit.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.
* ALT, alkaline phosphatase and bilirubin <=1x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* White blood cell count and absolute neutrophil count in the normal range.

Exclusion Criteria

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of clinically significant cardiovascular disease including

  * Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): male subjects with heart rate <45 and >100 beats per minute (bpm) and female subjects with heart rate <50 and >100 bpm, QRS duration (males and females) >120 millisecond (msec), QTc corrected by Fridericia's formula (QTcF) >450 msec for males and females.
  * Evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization).
  * History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
  * Conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree (type II) or higher], Wolf Parkinson White [WPW] syndrome) which in the opinion of the principal Investigator and Viiv Medical Monitor, will interfere with the safety for the individual subject.
  * Sinus pauses >3 seconds.
  * Any significant arrhythmia which, in the opinion of the principal Investigator and ViiV Medical Monitor, will interfere with the safety for the individual subject.
  * Non-sustained (>=3 consecutive ventricular ectopic beats) or sustained ventricular tachycardia.
* History of inflammatory bowel disease.
* History of cholecystectomy or other gastrointestinal surgery (except appendectomy more than three months prior to study).
* History of peptic ulceration or pancreatitis within the preceding 6 months of screening.
* Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrolment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrolment.
* Current or past history of uveitis.
* Any other medical condition which, in the judgment of the investigator and medical monitor, could jeopardize the safety of the subject or the integrity of the data derived from that subject. This includes but is not limited to any pre-existing condition that interferes with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drug.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and ViiV Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks. One drink is equivalent to 12 gram of alcohol, 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* A history of regular use of tobacco, or nicotine-containing products within 30 days prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of Hepatitis B surface antigen (HBsAg) positivity at screening or within 3 months prior to first dose of study treatment. Positive Hepatitis B core antibody (HBcAb) with negative hepatitis B surface antibody should also be excluded.
* Positive Hepatitis C antibody test.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* A positive QuantiFERON Gold test or clinical evidence of tuberculosis (TB) infection.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20363

REFERENCES:
- [Background] Ford SL, Lou Y, Lewis N, Kostapanos M, D'Amico R, Spreen W, Patel P. Effect of rifabutin on the pharmacokinetics of oral cabotegravir in healthy subjects. Antivir Ther. 2019;24(4):301-308. doi: 10.3851/IMP3306. PMID 30896438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 participants were enrolled from one center in the United Kingdom. The study was conducted from 06 June 2017 to 07 September 2017.
Pre-assignment Details: A total of 26 participants were screened for the study. Of these, 6 participants did not meet the inclusion/exclusion criteria and 5 participants (reserved participants) were eligible however they did not participate in the study. Therefore, 15 participants were enrolled and received at least one dose of study medication.
Groups:
- CAB 30 mg Followed by RBT 300 mg + CAB 30 mg: Eligible participants received cabotegravir (CAB) 30 milligrams (mg) oral tablets once daily for 14 days (Day 1 to Day 14) during Period 1 and rifabutin (RBT) 300 mg (2x150 mg) oral capsules once daily along with CAB 30 mg oral tablets once daily for 14 days (Day 15 to Day 28) during Period 2.
Period: Period 1 (Day 1 to Day 14)
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Started | 15
Completed | 14
Not Completed | 1
Not completed — Protocol-Defined Stopping criteria | 1
Period: Period 2 (Day 15 to Day 28)
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Started | 14
Completed | 12
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- CAB 30 mg Followed by RBT 300 mg + CAB 30 mg: Eligible participants received CAB 30 mg oral tablets once daily for 14 days (Day 1 to Day 14) during Period 1 and RBT 300 mg (2x150 mg) oral capsules once daily along with CAB 30 mg oral tablets once daily for 14 days (Day 15 to Day 28) during Period 2.
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 1
  White - White/Caucasian/European | 14

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Plasma CAB Pharmacokinetic (PK) Parameter: Area Under the Concentration-time Curve Over One Dosing Interval (AUC [0 to Tau])
Description: Blood samples for PK analysis of CAB were collected at pre-dose (within 15 minutes prior to dose) on Days 13 and 14; and 1, 2, 3, 4, 8, 12, and 24 hours post-dose on Day 14, pre-dose (within 15 minutes prior to dose) on Days 26, 27 and 28; and 1, 2, 3, 4, 8, 12 and 24 hours post-dose on Day 28. AUC (0 to tau) was calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. PK Summary Population included participants who had CAB PK parameter estimates from both serial PK sampling time periods 1 and 2. Comparisons were made for the repeated dose PK parameters of CAB when given alone in Period 1 and when co-administered with steady-state RBT in Period 2.
Time Frame: Pre-dose (within 15 minutes prior to dose) on Days 13 and 14; and 1, 2, 3, 4, 8, 12, and 24 hours post-dose on Day 14, pre-dose (within 15 minutes prior to dose) on Days 26, 27 and 28; and 1, 2, 3, 4, 8, 12 and 24 hours post-dose on Day 28
Population: PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram * hour per milliliter
Groups:
- CAB 30 mg: Eligible participants received CAB 30 mg oral tablets once daily for 14 days (Day 1 to Day 14) during Period 1.
- RBT 300 mg + CAB 30 mg: Eligible participants received RBT 300 mg (2x150 mg) oral capsules once daily along with CAB 30 mg oral tablets once daily for 14 days (Day 15 to Day 28) during Period 2.
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 12 | 12
Microgram * hour per milliliter | 103.978 (28.3) | 81.715 (29.9)
Statistical Analysis 1: Comparison: CAB 30 mg vs RBT 300 mg + CAB 30 mg; Test type: Other; Ratio = 0.786, 90% CI 2-sided [0.743 to 0.831]

2. Primary Outcome: Assessment of Plasma CAB PK Parameter: Maximum Observed Concentration (Cmax)
Description: Blood samples for PK analysis of CAB were collected at pre-dose (within 15 minutes prior to dose) on Days 13 and 14; and 1, 2, 3, 4, 8, 12, and 24 hours post-dose on Day 14, pre-dose (within 15 minutes prior to dose) on Days 26, 27 and 28; and 1, 2, 3, 4, 8, 12 and 24 hours post-dose on Day 28. Cmax was determined directly from the concentration-time data. Comparisons were made for the repeated dose PK parameters of CAB when given alone in Period 1 and when co-administered with steady-state RBT in Period 2.
Time Frame: as for outcome 1
Population: PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 12 | 12
Micrograms per milliliter | 6.356 (24.7) | 5.246 (24.3)
Statistical Analysis 1: Comparison: CAB 30 mg vs RBT 300 mg + CAB 30 mg; Test type: Other; Ratio = 0.825, 90% CI 2-sided [0.761 to 0.895]

3. Secondary Outcome: Assessment of Plasma CAB PK Parameter: Concentration at the End of the Dosing Interval (Ctau)
Description: Blood samples for PK analysis of CAB were collected at pre-dose (within 15 minutes prior to dose) on Days 13 and 14; and 1, 2, 3, 4, 8, 12, and 24 hours post-dose on Day 14, pre-dose (within 15 minutes prior to dose) on Days 26, 27 and 28; and 1, 2, 3, 4, 8, 12 and 24 hours post-dose on Day 28. Comparisons were made for the repeated dose PK parameters of CAB when given alone in Period 1 and when co-administered with steady-state RBT in Period 2.
Time Frame: as for outcome 1
Population: PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 12 | 12
Micrograms per milliliter | 3.359 (34.3) | 2.479 (36.3)
Statistical Analysis 1: Comparison: CAB 30 mg vs RBT 300 mg + CAB 30 mg; Test type: Other; Ratio = 0.738, 90% CI 2-sided [0.702 to 0.776]

4. Secondary Outcome: Assessment of Plasma CAB PK Parameter: Time of Occurrence of Cmax (Tmax)
Description: Blood samples for PK analysis of CAB were collected at pre-dose (within 15 minutes prior to dose) on Days 13 and 14; and 1, 2, 3, 4, 8, 12, and 24 hours post-dose on Day 14, pre-dose (within 15 minutes prior to dose) on Days 26, 27 and 28; and 1, 2, 3, 4, 8, 12 and 24 hours post-dose on Day 28. Tmax was determined directly from the concentration-time data.
Time Frame: as for outcome 1
Population: PK Summary Population
Measure: Median (Full Range); unit: Hours
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 12 | 12
Hours | 3.000 [1.00 to 4.00] | 2.500 [1.00 to 4.00]

5. Secondary Outcome: Assessment of Plasma CAB PK Parameter: Terminal Phase Half-life (t1/2)
Description: Blood samples for PK analysis of CAB were collected at pre-dose (within 15 minutes prior to dose) on Days 13 and 14; and 1, 2, 3, 4, 8, 12, and 24 hours post-dose on Day 14, pre-dose (within 15 minutes prior to dose) on Days 26, 27 and 28; and 1, 2, 3, 4, 8, 12 and 24 hours post-dose on Day 28. Apparent terminal half-life was calculated as: t1/2 = ln2 / Lambda_z, where Lambda_z is the terminal phase rate constant. Plasma t1/2 was not estimated for either period due to limited PK sampling in the terminal phase.
Time Frame: as for outcome 1
Population: PK Summary Population. Plasma t1/2 was not estimated for either period due to limited PK sampling in the terminal phase.
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Assessment of Plasma CAB PK Parameter: The Apparent Oral Clearance (CL/F)
Description: Blood samples for PK analysis of CAB were collected at pre-dose (within 15 minutes prior to dose) on Days 13 and 14; and 1, 2, 3, 4, 8, 12, and 24 hours post-dose on Day 14, pre-dose (within 15 minutes prior to dose) on Days 26, 27 and 28; and 1, 2, 3, 4, 8, 12 and 24 hours post-dose on Day 28. CL/F was calculated as CL/F =Dose/AUC(0 to tau).
Time Frame: as for outcome 1
Population: PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 12 | 12
Liters per hour | 0.289 (28.3) | 0.367 (29.9)
Statistical Analysis 1: Comparison: CAB 30 mg vs RBT 300 mg + CAB 30 mg; Test type: Other; Ratio = 1.272, 90% CI 2-sided [1.204 to 1.345]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect and associated with liver injury and impaired liver function. Safety Population comprised of all participants who enrolled in the study and received at least one dose of study drug.
Time Frame: Up to 10 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15 | 14
Participants
  Any AEs | 1 | 7
  Any SAEs | 0 | 1

8. Secondary Outcome: Concurrent Medication Assessment in Treatment Period 1 and 2
Description: Concurrent medications included paracetamol and ibuprofen. Number of participants who took concurrent medications during the study are presented.
Time Frame: Up to 10 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15 | 14
Participants
  Paracetamol | 0 | 3
  Ibuprofen | 0 | 1

9. Secondary Outcome: Assessment of Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Blood samples for hematology assessment were collected for basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
10^9 cells/Liter
  Basophils, Day -1, n=15 | 0.025 (0.0119)
  Basophils, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Basophils, On-treatment, Period 1 Day 13, n=14 | 0.031 (0.0141)
  Basophils, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Basophils, On-treatment, Period 2 Day 21, n=13 | 0.028 (0.0124)
  Basophils, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Basophils, On-treatment, Period 2 Day 27, n=12 | 0.018 (0.0106)
  Basophils, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Basophils, Follow-up, Period 1 Day 13, n=1 | 0.030 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Basophils, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Basophils, Follow-up, Period 2 Day 21, n=1 | 0.010 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Basophils, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Basophils, Follow-up, Period 2 Day 27, n=1 | 0.010 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Basophils, Follow-up, n=15 | 0.023 (0.0098)
  Eosinophils, On-treatment, Day -1, n=15 | 0.259 (0.2001)
  Eosinophils, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Eosinophils, On-treatment, Period 1 Day 13, n=14 | 0.285 (0.2264)
  Eosinophils, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Eosinophils, On-treatment, Period 2 Day 21, n=13 | 0.315 (0.2306)
  Eosinophils, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Eosinophils, On-treatment, Period 2 Day 27, n=12 | 0.219 (0.2815)
  Eosinophils, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Eosinophils, Follow-up, Period 1 Day 13, n=1 | 0.370 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Eosinophils, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Eosinophils, Follow-up, Period 2 Day 21, n=1 | 0.010 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Eosinophils, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Eosinophils, Follow-up, Period 2 Day 27, n=1 | 0.120 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Eosinophils, Follow-up, n=15 | 0.273 (0.2621)
  Lymphocytes, Day -1, n=15 | 2.509 (0.7383)
  Lymphocytes, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Lymphocytes, On-treatment, Period 1 Day 13, n=14 | 2.224 (0.6596)
  Lymphocytes, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Lymphocytes, On-treatment, Period 2 Day 21, n=13 | 2.071 (0.8625)
  Lymphocytes, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Lymphocytes, On-treatment, Period 2 Day 27, n=12 | 1.551 (0.6554)
  Lymphocytes, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Lymphocytes, Follow-up, Period 1 Day 13, n=1 | 1.200 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Lymphocytes, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Lymphocytes, Follow-up, Period 2 Day 21, n=1 | 0.310 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Lymphocytes, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Lymphocytes, Follow-up, Period 2 Day 27, n=1 | 0.480 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Lymphocytes, Follow-up, n=15 | 2.140 (0.7373)
  Monocytes, Day -1, n=15 | 0.561 (0.1570)
  Monocytes, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Monocytes, On-treatment, Period 1 Day 13, n=14 | 0.548 (0.1397)
  Monocytes, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Monocytes, On-treatment, Period 2 Day 21, n=13 | 0.628 (0.1579)
  Monocytes, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Monocytes, On-treatment, Period 2 Day 27, n=12 | 0.488 (0.1442)
  Monocytes, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Monocytes, Follow-up, Period 1 Day 13, n=1 | 0.360 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Monocytes, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Monocytes, Follow-up, Period 2 Day 21, n=1 | 0.480 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Monocytes, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Monocytes, Follow-up, Period 2 Day 27, n=1 | 0.790 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Monocytes, Follow-up, n=15 | 0.545 (0.1503)
  Neutrophils, Day -1, n=15 | 4.279 (1.2269)
  Neutrophils, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Neutrophils, On-treatment, Period 1 Day 13, n=14 | 3.306 (0.9964)
  Neutrophils, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Neutrophils, On-treatment, Period 2 Day 21, n=13 | 2.818 (1.0823)
  Neutrophils, On-treatment, Period 2 Day 21, n=12: number analyzed (Participants) | 12
  Neutrophils, On-treatment, Period 2 Day 21, n=12 | 1.979 (0.6006)
  Neutrophils, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Neutrophils, Follow-up, Period 1 Day 13, n=1 | 2.340 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Neutrophils, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Neutrophils, Follow-up, Period 2 Day 21, n=1 | 3.830 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Neutrophils, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Neutrophils, Follow-up, Period 2 Day 27, n=1 | 3.970 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Neutrophils, Follow-up, n=15 | 2.840 (0.8665)
  Platelets, Day -1, n=15 | 234.7 (34.58)
  Platelets, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Platelets, On-treatment, Period 1 Day 13, n=14 | 210.7 (31.46)
  Platelets, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Platelets, On-treatment, Period 2 Day 21, n=13 | 214.5 (31.04)
  Platelets, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Platelets, On-treatment, Period 2 Day 27, n=12 | 193.9 (34.47)
  Platelets, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Platelets, Follow-up, Period 1 Day 13, n=1 | 206.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Platelets, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Platelets, Follow-up, Period 2 Day 21, n=1 | 206.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Platelets, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Platelets, Follow-up, Period 2 Day 27, n=1 | 169.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Platelets, Follow-up, n=15 | 229.8 (45.57)
  Leukocytes, Day -1, n=15 | 7.633 (1.6572)
  Leukocytes, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Leukocytes, On-treatment, Period 1 Day 13, n=14 | 6.394 (1.5268)
  Leukocytes, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Leukocytes, On-treatment, Period 2 Day 21, n=13 | 5.859 (1.5835)
  Leukocytes, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Leukocytes, On-treatment, Period 2 Day 27, n=12 | 4.256 (1.3035)
  Leukocytes, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Leukocytes, Follow-up, Period 1 Day 13, n=1 | 4.300 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Leukocytes, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Leukocytes, Follow-up, Period 2 Day 21, n=1 | 4.640 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Leukocytes, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Leukocytes, Follow-up, Period 2 Day 27, n=1 | 5.370 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Leukocytes, Follow-up, n=15 | 5.822 (1.3583)

10. Secondary Outcome: Assessment of Hematology Parameters: Hematocrit and Reticulocytes/Erythrocytes (R/E)
Description: Blood samples for hematology assessment were collected for Hematocrit and R/E. NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Proportion of red blood cells in blood
  Hematocrit, Day -1, n=15 | 0.411 (0.02107)
  Hematocrit, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Hematocrit, On-treatment, Period 1 Day 13, n=14 | 0.427 (0.02432)
  Hematocrit, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Hematocrit, On-treatment, Period 2 Day 21, n=13 | 0.415 (0.02277)
  Hematocrit, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Hematocrit, On-treatment, Period 2 Day 27, n=12 | 0.425 (0.02139)
  Hematocrit, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Hematocrit, Follow-up, Period 1 Day 13, n=1 | 0.413 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Hematocrit, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Hematocrit, Follow-up, Period 2 Day 21, n=1 | 0.419 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Hematocrit, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Hematocrit, Follow-up, Period 2 Day 27, n=1 | 0.412 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Hematocrit, Follow-up, n=15 | 0.411 (0.01766)
  R/E, Day -1, n=15 | 0.008 (0.00228)
  R/E, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  R/E, On-treatment, Period 1 Day 13, n=14 | 0.008 (0.00248)
  R/E, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  R/E, On-treatment, Period 2 Day 21, n=13 | 0.008 (0.00209)
  R/E, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  R/E, On-treatment, Period 2 Day 27, n=12 | 0.006 (0.00219)
  R/E, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  R/E, Follow-up, Period 1 Day 13, n=1 | 0.013 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  R/E, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  R/E, Follow-up, Period 2 Day 21, n=1 | 0.009 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  R/E, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  R/E, Follow-up, Period 2 Day 27, n=1 | 0.003 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  R/E, Follow-up, n=15 | 0.010 (0.00270)

11. Secondary Outcome: Assessment of Hematology Parameter: Hemoglobin
Description: Blood samples for hematology assessment was collected for Hemoglobin. NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Grams per Liter
  Day -1, n=15 | 144.7 (7.25)
  Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Period 1 Day 13, n=14 | 143.5 (7.51)
  Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Period 2 Day 21, n=13 | 146.4 (8.13)
  Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Period 2 Day 27, n=12 | 144.2 (9.93)
  Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Follow-up, Period 1 Day 13, n=1 | 137.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 21, n=1 | 147.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 27, n=1 | 146.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, n=15 | 140.1 (6.04)

12. Secondary Outcome: Assessment of Hematology Parameter: Eryrocyte Mean Corpuscular Hemoglobin
Description: Blood samples for hematology assessment was collected for Eryrocyte Mean Corpuscular Hemoglobin. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Picograms
  Day -1, n=15 | 29.77 (1.457)
  On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  On-treatment, Period 1 Day 13, n=14 | 29.54 (1.536)
  On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  On-treatment, Period 2 Day 21, n=13 | 30.13 (1.329)
  On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  On-treatment, Period 2 Day 27, n=12 | 29.74 (1.466)
  Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Follow-up, Period 1 Day 13, n=1 | 29.30 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 21, n=1 | 27.80 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 27, n=1 | 30.90 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, n=15 | 29.49 (1.451)

13. Secondary Outcome: Assessment of Hematology Parameter: Erythrocye Mean Corpuscular Volume
Description: Blood samples for hematology assessment was collected for Erythrocyte Mean Corpuscular Volume. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Femtoliters
  Day -1, n=15 | 84.60 (3.522)
  On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  On-treatment, Period 1 Day 13, n=14 | 87.94 (2.829)
  On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  On-treatment, Period 2 Day 21, n=13 | 85.39 (3.367)
  On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  On-treatment, Period 2 Day 27, n=12 | 87.73 (3.997)
  Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Follow-up, Period 1 Day 13, n=1 | 88.20 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 21, n=1 | 79.20 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 27, n=1 | 87.10 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, n=15 | 86.59 (3.618)

14. Secondary Outcome: Assessment of Hematology Parameters: Erythrocytes and Reticulocytes
Description: Blood samples for hematology assessment were collected for Erythrocytes and reticulocytes. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
10^12 cells/Liter
  Erythrocytes, Day -1, n=15 | 4.870 (0.3068)
  Erythrocytes, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Erythrocytes, On-treatment, Period 1 Day 13, n=14 | 4.869 (0.3400)
  Erythrocytes, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Erythrocytes, On-treatment, Period 2 Day 21, n=13 | 4.868 (0.3173)
  Erythrocytes, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Erythrocytes, On-treatment, Period 2 Day 27, n=12 | 4.855 (0.3605)
  Erythrocytes, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Erythrocytes, Follow-up, Period 1 Day 13, n=1 | 4.680 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Erythrocytes, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Erythrocytes, Follow-up, Period 2 Day 21, n=1 | 5.290 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Erythrocytes, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Erythrocytes, Follow-up, Period 2 Day 27, n=1 | 4.730 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Erythrocytes, Follow-up, n=15 | 4.761 (0.3372)
  Reticulocytes, Day -1, n=15 | 0.043 (0.01246)
  Reticulocytes, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Reticulocytes, On-treatment, Period 1 Day 13, n=14 | 0.040 (0.01350)
  Reticulocytes, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Reticulocytes, On-treatment, Period 2 Day 21, n=13 | 0.040 (0.01097)
  Reticulocytes, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Reticulocytes, On-treatment, Period 2 Day 27, n=12 | 0.028 (0.00997)
  Reticulocytes, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Reticulocytes, Follow-up, Period 1 Day 13, n=1 | 0.064 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Reticulocytes, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Reticulocytes, Follow-up, Period 2 Day 21, n=1 | 0.051 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Reticulocytes, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Reticulocytes, Follow-up, Period 2 Day 27, n=1 | 0.014 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Reticulocytes, Follow-up, n=15 | 0.049 (0.01415)

15. Secondary Outcome: Assessment of Hematology Parameters: Erythrocytes Distribution Width (EDW)
Description: Blood samples for hematology assessment was collected for EDW. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Percentage of EDW
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Percentage of EDW
  Day -1, n=15 | 12.91 (0.513)
  On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  On-treatment, Period 1 Day 13, n=14 | 13.13 (0.595)
  On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  On-treatment, Period 2 Day 21, n=13 | 12.89 (0.641)
  On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  On-treatment, Period 2 Day 27, n=12 | 12.90 (0.624)
  Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Follow-up, Period 1 Day 13, n=1 | 13.40 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 21, n=1 | 13.60 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 27, n=1 | 12.40 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, n=15 | 12.90 (0.535)

16. Secondary Outcome: Assessment of Clinical Chemistry Parameters: Albumin and Protein
Description: Samples for clinical chemistry assessment were collected for Albumin and Protein. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Grams per Liter
  Albumin, Day -1, n=15 | 45.2 (1.90)
  Albumin, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Albumin, On-treatment, Period 1 Day 13, n=14 | 44.2 (2.58)
  Albumin, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Albumin, On-treatment, Period 2 Day 21, n=13 | 43.4 (2.06)
  Albumin, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Albumin, On-treatment, Period 2 Day 27, n=12 | 43.7 (1.87)
  Albumin, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Albumin, Follow-up, Period 1 Day 13, n=1 | 38.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Albumin, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Albumin, Follow-up, Period 2 Day 21, n=1 | 44.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Albumin, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Albumin, Follow-up, Period 2 Day 27, n=1 | 42.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Albumin, Follow-up, n=15 | 42.7 (1.59)
  Protein, Day -1, n=15 | 67.9 (3.98)
  Protein, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Protein, On-treatment, Period 1 Day 13, n=14 | 67.3 (3.22)
  Protein, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Protein, On-treatment, Period 2 Day 21, n=13 | 65.1 (3.82)
  Protein, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Protein, On-treatment, Period 2 Day 27, n=12 | 65.8 (4.00)
  Protein, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Protein, Follow-up, Period 1 Day 13, n=1 | 60.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Protein, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Protein, Follow-up, Period 2 Day 21, n=1 | 63.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Protein, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Protein, Follow-up, Period 2 Day 27, n=1 | 70.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Protein, Follow-up, n=15 | 63.7 (2.55)

17. Secondary Outcome: Assessment of Clinical Chemistry Parameters: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase (CK) and Gamma Glutamyl Transferase (GGT)
Description: Samples for clinical chemistry assessment were collected for ALP, AST, ALT, CK and GGT. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
International units per Liter
  ALP, Day -1, n=15 | 62.7 (14.52)
  ALP, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  ALP, On-treatment, Period 1 Day 13, n=14 | 60.1 (14.34)
  ALP, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  ALP, On-treatment, Period 2 Day 21, n=13 | 60.7 (13.94)
  ALP, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  ALP, On-treatment, Period 2 Day 27, n=12 | 59.9 (17.83)
  ALP, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  ALP, Follow-up, Period 1 Day 13, n=1 | 51.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  ALP, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  ALP, Follow-up, Period 2 Day 21, n=1 | 61.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  ALP, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  ALP, Follow-up, Period 2 Day 27, n=1 | 56.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  ALP, Follow-up, n=15 | 60.7 (13.35)
  ALT, Day -1, n=15 | 23.5 (7.07)
  ALT, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  ALT, On-treatment, Period 1 Day 13, n=14 | 25.5 (8.83)
  ALT, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  ALT, On-treatment, Period 2 Day 21, n=13 | 30.2 (20.12)
  ALT, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  ALT, On-treatment, Period 2 Day 27, n=12 | 30.8 (29.65)
  ALT, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  ALT, Follow-up, Period 1 Day 13, n=1 | 155.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  ALT, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  ALT, Follow-up, Period 2 Day 21, n=1 | 39.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  ALT, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  ALT, Follow-up, Period 2 Day 27, n=1 | 34.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  ALT, Follow-up, n=15 | 37.3 (23.40)
  AST, Day -1, n=15 | 18.5 (3.62)
  AST, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  AST, On-treatment, Period 1 Day 13, n=14 | 20.7 (6.85)
  AST, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  AST, On-treatment, Period 2 Day 21, n=13 | 20.9 (5.87)
  AST, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  AST, On-treatment, Period 2 Day 27, n=12 | 23.3 (11.48)
  AST, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  AST, Follow-up, Period 1 Day 13, n=1 | 83.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  AST, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  AST, Follow-up, Period 2 Day 21, n=1 | 26.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  AST, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  AST, Follow-up, Period 2 Day 27, n=1 | 37.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  AST, Follow-up, n=15 | 24.9 (9.44)
  CK, Day -1, n=15 | 133.6 (40.31)
  CK, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  CK, On-treatment, Period 1 Day 13, n=14 | 227.1 (303.97)
  CK, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  CK, On-treatment, Period 2 Day 21, n=13 | 104.2 (43.44)
  CK, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  CK, On-treatment, Period 2 Day 27, n=12 | 88.7 (42.09)
  CK, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  CK, Follow-up, Period 1 Day 13, n=1 | 1278.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  CK, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  CK, Follow-up, Period 2 Day 21, n=1 | 177.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  CK, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  CK, Follow-up, Period 2 Day 27, n=1 | 164.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  CK, Follow-up, n=15 | 144.3 (80.81)
  GGT, Day -1, n=15 | 25.5 (14.97)
  GGT, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  GGT, On-treatment, Period 1 Day 13, n=14 | 22.6 (13.20)
  GGT, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  GGT, On-treatment, Period 2 Day 21, n=13 | 26.8 (23.95)
  GGT, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  GGT, On-treatment, Period 2 Day 27, n=12 | 28.1 (28.25)
  GGT, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  GGT, Follow-up, Period 1 Day 13, n=1 | 17.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  GGT, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  GGT, Follow-up, Period 2 Day 21, n=1 | 36.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  GGT, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  GGT, Follow-up, Period 2 Day 27, n=1 | 82.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  GGT, Follow-up, n=15 | 36.1 (33.77)

18. Secondary Outcome: Assessment of Clinical Chemistry Parameters: Direct Bilirubin (DB), Bilirubin and Creatinine
Description: Samples for clinical chemistry assessment were collected for DB, bilirubin and creatinine. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Micromoles per Liter
  DB, Day -1, n=15 | 3.5 (2.00)
  DB, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  DB, On-treatment, Period 1 Day 13, n=14 | 3.5 (1.83)
  DB, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  DB, On-treatment, Period 2 Day 21, n=13 | 2.4 (1.45)
  DB, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  DB, On-treatment, Period 2 Day 27, n=12 | 2.2 (1.19)
  DB, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  DB, Follow-up, Period 1 Day 13, n=1 | 4.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  DB, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  DB, Follow-up, Period 2 Day 21, n=1 | 1.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  DB, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  DB, Follow-up, Period 2 Day 27, n=1 | 2.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  DB, Follow-up, n=15 | 2.9 (1.39)
  Bilirubin, Day -1, n=15 | 9.8 (6.72)
  Bilirubin, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Bilirubin, On-treatment, Period 1 Day 13, n=14 | 10.1 (5.83)
  Bilirubin, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Bilirubin, On-treatment, Period 2 Day 21, n=13 | 6.6 (4.74)
  Bilirubin, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Bilirubin, On-treatment, Period 2 Day 27, n=12 | 5.3 (2.99)
  Bilirubin, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Bilirubin, Follow-up, Period 1 Day 13, n=1 | 10.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Bilirubin, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Bilirubin, Follow-up, Period 2 Day 21, n=1 | 3.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Bilirubin, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Bilirubin, Follow-up, Period 2 Day 27, n=1 | 5.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Bilirubin, Follow-up, n=15 | 7.9 (3.83)
  Creatinine, Day -1, n=15 | 83.1 (7.71)
  Creatinine, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Creatinine, On-treatment, Period 1 Day 13, n=14 | 85.9 (11.02)
  Creatinine, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Creatinine, On-treatment, Period 2 Day 21, n=13 | 88.4 (9.43)
  Creatinine, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Creatinine, On-treatment, Period 2 Day 27, n=12 | 83.8 (10.69)
  Creatinine, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Creatinine, Follow-up, Period 1 Day 13, n=1 | 64.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Creatinine, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Creatinine, Follow-up, Period 2 Day 21, n=1 | 71.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Creatinine, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Creatinine, Follow-up, Period 2 Day 27, n=1 | 91.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Creatinine, Follow-up, n=15 | 80.7 (9.65)

19. Secondary Outcome: Assessment of Clinical Chemistry Parameters: Calcium, Chloride, Carbon Dioxide, Glucose, Potassium, Sodium and Urea
Description: Samples for clinical chemistry assessment were collected for Calcium, Chloride, Carbon Dioxide, Glucose, Potassium, Sodium and Urea. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Millimoles per Liter
  Calcium, Day -1, n=15 | 2.31 (0.0539)
  Calcium, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Calcium, On-treatment, Period 1 Day 13, n=14 | 2.34 (0.0770)
  Calcium, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Calcium, On-treatment, Period 2 Day 21, n=13 | 2.29 (0.0720)
  Calcium, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Calcium, On-treatment, Period 2 Day 27, n=12 | 2.28 (0.0844)
  Calcium, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Calcium, Follow-up, Period 1 Day 13, n=1 | 2.27 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Calcium, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Calcium, Follow-up, Period 2 Day 21, n=1 | 2.38 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Calcium, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Calcium, Follow-up, Period 2 Day 27, n=1 | 2.06 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Calcium, Follow-up, n=15 | 2.28 (0.0400)
  Chloride, Day -1, n=15 | 101.0 (1.73)
  Chloride, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Chloride, On-treatment, Period 1 Day 13, n=14 | 100.5 (1.45)
  Chloride, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Chloride, On-treatment, Period 2 Day 21, n=13 | 101.1 (2.40)
  Chloride, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Chloride, On-treatment, Period 2 Day 27, n=12 | 101.8 (2.14)
  Chloride, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Chloride, Follow-up, Period 1 Day 13, n=1 | 101.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Chloride, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Chloride, Follow-up, Period 2 Day 21, n=1 | 100.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Chloride, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Chloride, Follow-up, Period 2 Day 27, n=1 | 99.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Chloride, Follow-up, n=15 | 102.5 (2.07)
  Carbon Dioxide, Day -1, n=15 | 25.6 (1.12)
  Carbon Dioxide, On-treatment, Period 1 Day13, n=14: number analyzed (Participants) | 14
  Carbon Dioxide, On-treatment, Period 1 Day13, n=14 | 25.3 (1.38)
  Carbon Dioxide, On-treatment, Period 2 Day21, n=13: number analyzed (Participants) | 13
  Carbon Dioxide, On-treatment, Period 2 Day21, n=13 | 27.4 (2.10)
  Carbon Dioxide, On-treatment, Period 2 Day27, n=12: number analyzed (Participants) | 12
  Carbon Dioxide, On-treatment, Period 2 Day27, n=12 | 24.7 (3.11)
  Carbon Dioxide, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Carbon Dioxide, Follow-up, Period 1 Day 13, n=1 | 25.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Carbon Dioxide, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Carbon Dioxide, Follow-up, Period 2 Day 21, n=1 | 27.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Carbon Dioxide, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Carbon Dioxide, Follow-up, Period 2 Day 27, n=1 | 20.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Carbon Dioxide, Follow-up, n=15 | 25.7 (1.76)
  Glucose, Day -1, n=15 | 5.27 (1.077)
  Glucose, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Glucose, On-treatment, Period 1 Day 13, n=14 | 5.51 (0.487)
  Glucose, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Glucose, On-treatment, Period 2 Day 21, n=13 | 5.45 (0.399)
  Glucose, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Glucose, On-treatment, Period 2 Day 27, n=12 | 5.95 (1.103)
  Glucose, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Glucose, Follow-up, Period 1 Day 13, n=1 | 5.00 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Glucose, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Glucose, Follow-up, Period 2 Day 21, n=1 | 5.40 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Glucose, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Glucose, Follow-up, Period 2 Day 27, n=1 | 6.00 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Glucose, Follow-up, n=15 | 5.35 (0.374)
  Potassium, Day -1, n=15 | 4.22 (0.166)
  Potassium, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Potassium, On-treatment, Period 1 Day 13, n=14 | 4.29 (0.250)
  Potassium, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Potassium, On-treatment, Period 2 Day 21, n=13 | 4.36 (0.386)
  Potassium, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Potassium, On-treatment, Period 2 Day 27, n=12 | 4.29 (0.247)
  Potassium, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Potassium, Follow-up, Period 1 Day 13, n=1 | 3.90 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Potassium, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Potassium, Follow-up, Period 2 Day 21, n=1 | 4.00 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Potassium, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Potassium, Follow-up, Period 2 Day 27, n=1 | 4.10 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Potassium, Follow-up, n=15 | 4.31 (0.183)
  Sodium, Day -1, n=15 | 141.1 (1.28)
  Sodium, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Sodium, On-treatment, Period 1 Day 13, n=14 | 139.6 (1.82)
  Sodium, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Sodium, On-treatment, Period 2 Day 21, n=13 | 140.3 (2.36)
  Sodium, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Sodium, On-treatment, Period 2 Day 27, n=12 | 139.8 (2.09)
  Sodium, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Sodium, Follow-up, Period 1 Day 13, n=1 | 139.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Sodium, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Sodium, Follow-up, Period 2 Day 21, n=1 | 140.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Sodium, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Sodium, Follow-up, Period 2 Day 27, n=1 | 137.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Sodium, Follow-up, n=15 | 141.1 (2.02)
  Urea, Day -1, n=15 | 5.73 (1.4048)
  Urea, On-treatment, Period 1 Day 13, n=14: number analyzed (Participants) | 14
  Urea, On-treatment, Period 1 Day 13, n=14 | 5.19 (1.0830)
  Urea, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  Urea, On-treatment, Period 2 Day 21, n=13 | 5.69 (1.3678)
  Urea, On-treatment, Period 2 Day 27, n=12: number analyzed (Participants) | 12
  Urea, On-treatment, Period 2 Day 27, n=12 | 5.18 (1.2104)
  Urea, Follow-up, Period 1 Day 13, n=1: number analyzed (Participants) | 1
  Urea, Follow-up, Period 1 Day 13, n=1 | 4.69 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Urea, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Urea, Follow-up, Period 2 Day 21, n=1 | 2.79 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Urea, Follow-up, Period 2 Day 27, n=1: number analyzed (Participants) | 1
  Urea, Follow-up, Period 2 Day 27, n=1 | 4.09 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Urea, Follow-up, n=15 | 5.34 (1.2189)

20. Secondary Outcome: Number of Participants With Abnormal Urinalysis Result
Description: Samples for urinalysis assessment was collected at Day -1, Day 13, Day 21, Day 27 and during follow-up period (10 to 14 daya after last dose). Data for participants with abnormal urinalysis results has been presented.
Time Frame: Day -1, Day 13, Day 21, Day 27 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15 | 14
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: ECG measurements was performed with the participant in a semi-supine position having rested in this position for at least 10 minutes beforehand. Data has been presented for Period 1, Day 14 pre-dose which showed abnormal- not clinically significant ECG finding. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day 1, 14, 21, 28 and follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 14 | 12
Participants | 1 | 0

22. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs measurement was done in semi-supine position after 10 minutes rest and included SBP and DBP. Two blood pressure measurement were taken at pre-dose on Day 1, at least 1 minute apart. The mean value recorded at pre-dose was classified as Baseline. Single blood pressure was obtained at all other time points during the study. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline to follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Millimeters of Mercury
  SBP, On-treatment, Period 1 Day 14, n=14: number analyzed (Participants) | 14
  SBP, On-treatment, Period 1 Day 14, n=14 | -2.5 (9.17)
  SBP, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  SBP, On-treatment, Period 2 Day 21, n=13 | 1.5 (11.90)
  SBP, On-treatment, Period 2 Day 28, n=12: number analyzed (Participants) | 12
  SBP, On-treatment, Period 2 Day 28, n=12 | 0.5 (8.74)
  SBP, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  SBP, Follow-up, Period 2 Day 21, n=1 | 17.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  SBP, Follow-up, n=15 | 3.7 (12.85)
  DBP, On-treatment, Period 1 Day 14, n=14: number analyzed (Participants) | 14
  DBP, On-treatment, Period 1 Day 14, n=14 | 0.8 (7.61)
  DBP, On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  DBP, On-treatment, Period 2 Day 21, n=13 | 2.0 (9.10)
  DBP, On-treatment, Period 2 Day 28, n=12: number analyzed (Participants) | 12
  DBP, On-treatment, Period 2 Day 28, n=12 | -1.6 (4.21)
  DBP, Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  DBP, Follow-up, Period 2 Day 21, n=1 | 9.5 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  DBP, Follow-up, n=15 | 3.3 (9.04)

23. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Vital signs measurement was done in semi-supine position after 10 minutes rest and included pulse rate. Two pulse rate measurement were taken at pre-dose on Day 1, at least 1 minute apart. The mean value recorded at pre-dose was classified as Baseline. Single pulse rate was obtained at all other time points during the study. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. NA indicated data not available since only one participant was analyzed, therefore standard deviation was not derived. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline to follow-up (10 to 14 days after last dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | CAB 30 mg Followed by RBT 300 mg + CAB 30 mg
Number analyzed (Participants) | 15
Beats/minute
  On-treatment, Period 1 Day 14, n=14: number analyzed (Participants) | 14
  On-treatment, Period 1 Day 14, n=14 | -4.5 (8.31)
  On-treatment, Period 2 Day 21, n=13: number analyzed (Participants) | 13
  On-treatment, Period 2 Day 21, n=13 | -6.2 (9.98)
  On-treatment, Period 2 Day 28, n=12: number analyzed (Participants) | 12
  On-treatment, Period 2 Day 28, n=12 | 3.4 (9.52)
  Follow-up, Period 2 Day 21, n=1: number analyzed (Participants) | 1
  Follow-up, Period 2 Day 21, n=1 | 39.0 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
  Follow-up, n=15 | -1.3 (10.58)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from start of the study up to follow-up (up to 10 weeks).
Description: AEs and SAEs were collected for the Safety Population which comprised of all participants who enrolled in the study and received at least one dose of study drug was included in the Safety Population.
Arm/Group | CAB 30 mg | RBT 300 mg + CAB 30 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/14
Other Adverse Events (participants affected / at risk) | 1/15 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAB 30 mg (N=15) | RBT 300 mg + CAB 30 mg (N=14)
Alanine aminotransferase increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CAB 30 mg (N=15) | RBT 300 mg + CAB 30 mg (N=14)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT03149848/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03149848/SAP_001.pdf